CLINICAL TRIAL: NCT04975074
Title: Prospective Study of Iron Deficiency Anemia in Twin Pregnancy
Brief Title: Iron Deficiency Anemia in Twin Pregnancies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caixia Liu, Clinical Professor, Shengjing Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IDA in TP
Record Dates: First submitted 2021-06-21; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Anemia, Iron-Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron; ferrous sulfate; ferrous succinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anemia Correction Group (Experimental): Continue to take the current medication orally at the current dose
  Interventions: Drug: Iron
- Anemia uncorrected group (Experimental): Continue to take the current medication orally at the current dose
  Interventions: Drug: Iron

INTERVENTIONS:
Drug: Iron — One of each type of iron was taken orally according to the instructions and followed every two weeks
  Other Names: ferrous sulfate; polyferose; ferrous succinate; Chinese medicine filling iron agent

SUMMARY:
All pregnant women with twin pregnancies were given oral iron according to the current recommended dose. Blood routine and ferritin were monitored during pregnancy to understand the therapeutic effect of oral iron on iron deficiency anemia and iron deficiency in pregnant women with twin pregnancies

DETAILED DESCRIPTION:
All pregnant women with twin pregnancies were given oral iron according to the current recommended dose. Blood routine and ferritin were monitored every 2-4 weeks during pregnancy to understand the therapeutic effect of oral iron on iron deficiency anemia and iron deficiency in pregnant women with twin pregnancies.After delivery, we will test the neonatal ferritin and hemoglobin status. Our aim was to investigate the effects of iron supplementation during twin pregnancy on maternal and neonatal ferritin and anemia.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* Pregnant women with twin pregnancies

Exclusion Criteria:

* Single pregnancy
* Types of anemia other than iron deficiency anemia

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Routine blood | 2-4 weeks after antenatal care
  Routine blood and serum ferritin（ng/ml）were checked 2-4 weeks

SECONDARY OUTCOMES:
serum ferritin | 2-4 weeks after antenatal care
  routine blood and serum ferritin（ng/ml）were checked 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caixia Liu, Study Chair — Shengjing Hospital of CMU

IPD SHARING:
Plan to Share IPD: No